CLINICAL TRIAL: NCT04830865
Title: Adaptation and Validation of Frailty Scales in Critically Ill Patients Admitted to Intensive Care Units in Spain
Brief Title: Adaptation and Validation of Frailty Scales in Intensive Care Units in Spain
Status: Completed | Type: Observational
Sponsor: Hospital Universitario Getafe (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Susana Arias Rivera, Principal Investigator, Hospital Universitario Getafe
Other Study IDs: PI20/01231; CEIM19/42 (Other: Hospital Universitario de Getafe)
Record Dates: First submitted 2021-03-25; First posted 2021-04-05 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Frailty Syndrome
Keywords: Frailty; critical care; gender; reliability; validity; study transcultural; quality of life
MeSH Terms: conditions — Frailty; Coitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Increased life expectancy leads to population aging, increased morbidities and aging of hospitalized patients. The acquisition of frailty leads to worse outcomes derived from hospitalization, but although frailty has been related to aging, young patients admitted to Intensive Care Units (ICU) with frailty have also been found to have worse outcomes than non-frail patients. This unfavorable evolution could be related to the acquisition of the post-uci syndrome (physical, mental and cognitive sequelae at discharge from the ICU), since high frailty scores favor this syndrome.

The use of frailty scales on admission to the ICU could provide early detection of patients most likely to develop post-ICU syndrome, regardless of age, and redirect our care to those who need it most. Some scales that measure frailty in elderly patients have been used in the ICU, but although they have been validated in their original language, they need to be adapted and validated in Spanish.

Objectives. Adaptation and validation of the Clinical Frailty Scale (CFS) and the FRAIL Scale in ICU patients of different ages, in women and in men.

Methodology. Study developed in two phases.Phase 1, adaptation to Spanish of the scales (translation, pilot, back-translation, correlation); Phase 2, analysis of their metric properties (Validity, Reliability, Sensitivity, Minimum important difference) by means of a multicenter observational study (7 ICUs in Spain), prospective, descriptive, of a cohort of critical patients with one-year follow-up (at 3, 6, 9 and 12 months after hospital discharge).

ELIGIBILITY:
Inclusion Criteria:

- Critical care patients over 18 years who have given their consent personally.

Exclusion Criteria:

* Patients admitted with a diagnosis of present or imminent brain death,
* readmissions previously included,
* patients whose expected stay is less than 48 hours
* patients with comunication problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who remain hospitalized for more than 48 hours in any of the 8 Spanish intensive care units participating in the study, they will be candidates for inclusion in the study.
Sampling Method: Non-Probability Sample
Enrollment: 512 (Actual)
Dates: Start 2019-09-15 (Actual); Primary Completion 2024-10-05 (Actual); Study Completion 2024-10-05 (Actual)

PRIMARY OUTCOMES:
Fragility scales's validation | 2 years
  100% scale sensitivity

SECONDARY OUTCOMES:
Obtaining adapted scales to patients in intensive care units in Spain | 6 months
  Through a process of cross-cultural, FRAIL scale will be implemented in spanish. Minimun value is 0 and maximum value is 5. Value of 0 is not frail, values of 1 or 2 is prefrail and values of 3 to 5 is frail.
Obtaining adapted scales to patients in intensive care units in Spain | 6 months
  Through a process of cross-cultural adaptation, Clinical Frailty Scale (CFS) will be implemented in spanish. Minimun value is 0 and maximum value is 9. Values of 0 to 3 is not frail, values of 4 is vulnerable, and 5 or 9 is frail.
Assessment of the predictive, convergent and divergent validity of the scales obtained (with respect to the original ones) | 2 years
  Using statistical tests, the validity of the scales will be estimated in relation to the variables which it should or should not have concordance and its predictive capacity.
Assessment of the interobserver and intraobserver reliability of the scales obtained (with respect to the original ones) | 2 years
  Through statistical tests, the interobserver and intraobserver concordance between nurses and physicians will be estimated.
Assessment of the sensitivity to change of the scales obtained (with respect to the original ones) | 1 year
  Through statistical tests, the floor and ceiling of the scales and the change in the score of the scales obtained between baseline and 3, 6, 9 and 12 months after hospital discharge will be assessed.
Assessment of the minimum important difference of the scales obtained | 2 years
  The relevance of the change in the score on the scales will be assessed, from the point of view of the patient and the professionals, related to quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario de Getafe, Getafe, Madrid, Spain